CLINICAL TRIAL: NCT01401439
Title: Longitudinal Assessment of Fat Free Mass Index and Its Impact on Lung Health and Overall Health Metrics in Pediatric Patients With Cystic Fibrosis
Brief Title: Assessment of Fat Free Mass Index and Its Impact on Health in Children With Cystic Fibrosis
Acronym: GAIA
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 131677
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; body mass index; fat free mass; Children with cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out whether measurement of body composition has a prognostic value on clinical and overall outcome in pediatric patients with cystic fibrosis.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is one of the most common life-threatening inherited disorders affecting 1/35000 individuals in the US. In the past decades, the median predicted survival of CF patients has increased significantly from 10-12 to over 37 years (1). One of the major factors contributing to increased survival has been the understanding of the role of optimal nutrition on overall health status of individuals with CF.

Forced expiratory volume in one second (FEV1) is currently the best predictor of pulmonary health in CF, and malnutrition in a person of any age with CF has a negative impact on lung function with a more rapid yearly decline in FEV1. Recent data from the Cystic Fibrosis Foundation (CFF) patient registries in the United States and Canada were analyzed to determine whether any association existed between pulmonary function as measured by FEV1 and Body mass index (BMI) for age. BMI-for-age percentile values >50th percentile were associated with well-preserved lung function and lower values of BMI were associated with incrementally lower values of FEV1 (2). Thus, the CFF recommended that children with CF between the ages of 2 and 20 years maintain a BMI a≥50th percentile for age and sex. However, several publications have demonstrated that fat free muscle (FFM) wasting is evident even in individuals with a BMI > 50th percentile, and it is unknown whether BMI percentile adequately reflects changes in body composition in this group of patients; therefore, BMI might not be the best marker indicating an optimal nutritional status.

Limitations of BMI as a marker of optimal Nutrition: fat mass versus muscle mass In individuals with CF, BMI is used to assess appropriateness of weight to height for age and sex. Since there is a strong association between BMI and overall health metrics, especially lung health, the CFF recommends that children with CF maintain a BMI ≥50th percentile for age and sex. However, an apparent loss of skeletal muscle may occur in CF patients who retain their normal body weight, indicating that BMI does not provide any information about body compartments and may fail to detect subtle alterations in body composition. Although several epidemiologic studies showed that CF patients who maintain BMI> 50th percentile will have improved lung functions and survival, recent data indicate that the preserved FFM instead of BMI may have an impact on overall survival in CF (7). Because of the variability in the levels of both fat mass and fat-free mass, and the many combinations of fat mass index and FFM index associated with the same BMI, this weight-height index needs to be carefully interpreted. Because high levels of BMI-for-age are associated with substantial increases in fat mass, BMI is most useful as a measure of obesity. In chronic inflammatory diseases, a change in regional fat distribution is observed with a shift to a more central fat distribution. The latter is associated with an increase in low-grade chronic inflammation, insulin resistance, and cardiovascular risk (8). Therefore, BMI is a good index for assessment of obesity in otherwise normal children, but not adequate or sufficient in the CF population.

In summary, some pediatric patients with CF may have a decreased Fat-free Mass Index (FFMI) with a well preserved BMI of ≥50th percentile. Conversely, some patient might have a BMI<50th percentile with normal FFMI associated with overall well-being. Current practice forces CF patients to consume high fat and caloric nutrients to maintain a BMI >50th percentiles incurring the costs of causing anxiety, stress, daily struggle in the family with a potential increase in the pro-inflammatory state due to central fat accumulation. The outcome of the proposed study will contribute to the understanding of the relationships between BMI, muscle wasting and markers of health and wellbeing. If our study demonstrates that a well maintained FFMI rather than the BMI correlates better with good health status in CF, it may result in changes of current nutrition practice in CF at the national or even international level.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who already have a diagnosis of CF based on universal diagnostic criteria
* Age 7 to 17 years at the time of enrollment
* Under routine medical control at the CF center of Arkansas Children's Hospital(ACH)
* Clinically stable in CF symptoms as determined by investigators

Exclusion Criteria:

* Unstable current diagnosis of metabolic diseases including liver (cirrhosis) or renal disease
* Failure to give informed consent
* Individuals with pacemakers
* Pregnancy in females of childbearing age. A pregnancy test will be performed on females who are post-menarche before performing a DEXA scan

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cystic fibrosis 7-17 years followed at Arkansas Children's hospital Cystic Fibrosis Care Center
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
body composition (bone mineral density) | change from baseline to 18 months
  Compare Dual Energy X-Ray Absorptiometry (DEXA) analysis to GAIA device

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Berlinski, MD, Principal Investigator — University of Arkansas for Medical Sciences/Arkansas Children's Hospital
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Zemel BS, Jawad AF, FitzSimmons S, Stallings VA. Longitudinal relationship among growth, nutritional status, and pulmonary function in children with cystic fibrosis: analysis of the Cystic Fibrosis Foundation National CF Patient Registry. J Pediatr. 2000 Sep;137(3):374-80. doi: 10.1067/mpd.2000.107891. PMID 10969263
- [Background] Ionescu AA, Evans WD, Pettit RJ, Nixon LS, Stone MD, Shale DJ. Hidden depletion of fat-free mass and bone mineral density in adults with cystic fibrosis. Chest. 2003 Dec;124(6):2220-8. doi: 10.1378/chest.124.6.2220. PMID 14665504
- [Background] Bolton CE, Ionescu AA, Evans WD, Pettit RJ, Shale DJ. Altered tissue distribution in adults with cystic fibrosis. Thorax. 2003 Oct;58(10):885-9. doi: 10.1136/thorax.58.10.885. PMID 14514945
- [Background] Wolfe RR. Regulation of muscle protein by amino acids. J Nutr. 2002 Oct;132(10):3219S-24S. doi: 10.1093/jn/131.10.3219S. PMID 12368421
- [Background] Reeds PJ, Fjeld CR, Jahoor F. Do the differences between the amino acid compositions of acute-phase and muscle proteins have a bearing on nitrogen loss in traumatic states? J Nutr. 1994 Jun;124(6):906-10. doi: 10.1093/jn/124.6.906. No abstract available. PMID 7515956
- [Background] Ionescu AA, Nixon LS, Evans WD, Stone MD, Lewis-Jenkins V, Chatham K, Shale DJ. Bone density, body composition, and inflammatory status in cystic fibrosis. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):789-94. doi: 10.1164/ajrccm.162.3.9910118. PMID 10988084
- [Background] Moriconi N, Kraenzlin M, Muller B, Keller U, Nusbaumer CP, Stohr S, Tamm M, Puder JJ. Body composition and adiponectin serum concentrations in adult patients with cystic fibrosis. J Clin Endocrinol Metab. 2006 Apr;91(4):1586-90. doi: 10.1210/jc.2005-2135. Epub 2006 Feb 7. PMID 16464949
- [Background] Engelen MP, Schols AM, Does JD, Wouters EF. Skeletal muscle weakness is associated with wasting of extremity fat-free mass but not with airflow obstruction in patients with chronic obstructive pulmonary disease. Am J Clin Nutr. 2000 Mar;71(3):733-8. doi: 10.1093/ajcn/71.3.733. PMID 10702166
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] Quittner AL, Sweeny S, Watrous M, Munzenberger P, Bearss K, Gibson Nitza A, Fisher LA, Henry B. Translation and linguistic validation of a disease-specific quality of life measure for cystic fibrosis. J Pediatr Psychol. 2000 Sep;25(6):403-14. doi: 10.1093/jpepsy/25.6.403. PMID 10980045